CLINICAL TRIAL: NCT04098614
Title: Barriers to Substance Use Disorder Recovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prisma Health-Upstate (Other)
Collaborators: Clemson University (Other); Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Prerana Roth, Clinical Assistant Professor, Prisma Health-Upstate
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00087080
Record Dates: First submitted 2019-06-11; First posted 2019-09-23 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2021-02

CONDITIONS: Substance Use Disorders
Keywords: recovery coaching; risk factors; substance abuse; EEG
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: The investigator/study personnel inform the participant regarding which arm they have been assigned and inform a recovery coach if the participant is randomized to the intervention arm.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Recovery Coach Intervention (Experimental): Experimental: Recovery Coach Intervention Participants randomized to the intervention arm are linked to a recovery peer coach while they are in the hospital. Recovery peer coaches are provided to the participant by Faces and Voices of Recovery (FAVOR)
  - Greenville. Recovery coaches are Certified Peer Support Specialists (CPSS), individuals who have firsthand experience in successful recovery and are trained in using recovery-oriented tools to help peers overcome addiction. FAVOR offers immediate access to a personal coach, a local center, and assistance to off-site intervention and recovery resources in the community. They provide twice weekly contact with participants.
  Interventions: Behavioral: Recovery Coach Intervention
- Standard of Care Control (No Intervention): Patients in the control condition receive the current standard of care, which entails a treatment referral with a list of addiction recovery facilities, groups, and resources. It is the patient's responsibility to call a treatment facility or group on the list and thus relies on self-referral. The medical team is not permitted to call a facility or group on behalf of the patient. The physician may counsel the patient on the dangers of substance abuse and addiction, but the extent of counseling is variable and dependent on the individual physician.

INTERVENTIONS:
Behavioral: Recovery Coach Intervention — Participants randomized to the intervention arm are linked to a recovery peer coach while they are in the hospital. Recovery peer coaches are provided to the participant by Faces and Voices of Recovery (FAVOR) - Greenville. Recovery coaches are Certified Peer Support Specialists (CPSS), individuals who have firsthand experience in successful recovery and are trained in using recovery-oriented tools to help peers overcome addiction. FAVOR offers immediate access to a personal coach, a local center, and assistance to off-site intervention and recovery resources in the community. They provide twice weekly contact with participants.
  Arms: Recovery Coach Intervention

SUMMARY:
The study purpose is to investigate how an inpatient recovery coaching intervention can overcome or mitigate specific risk factors and barriers to initiating and maintaining Substance Use Disorder recovery. This study will offer insight into how and why an inpatient link to recovery coaching is effective for promoting long-term Substance Use Disorder recovery.

DETAILED DESCRIPTION:
Substance Use Disorder (SUD) is a prevalent disease that impacts an estimated 24 million Americans each year. The life-altering consequences of SUD are both diverse and severe, influencing mortality, the workplace, and economics. The goal of this study is to determine how specific risk factors of relapse and barriers to recovery, including neurocognitive, health, personal, social, financial, and situational barriers, can be overcome or changed through a recovery coaching intervention. This work seeks to provide a mechanism to demonstrate exactly how and why this potential new model of care (recovery coaching) is effective, rather than simply assessing if it can work. To accomplish this aim, the change between baseline and 6-month assessments will be assessed. Then, the difference in the change between individuals assigned to the current standard of care and patients assigned to inpatient recovery will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 60
* English speaking;
* Identified by healthcare provider as having Substance Use Disorder
* Recent substance use
* Currently admitted to the Medical Teaching Services, general medicine hospitalist services, or Infectious Disease Consult service at Greenville Memorial Hospital

Exclusion Criteria:

* Are unable to provide informed consent (intubation, confusion, etc.) during hospitalization
* Are admitted for marijuana use only
* Are admitted for cocaine use only
* Are pregnant

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 99 (Actual)
Dates: Start 2019-09-03 (Actual); Primary Completion 2020-12-18 (Actual); Study Completion 2020-12-18 (Actual)

PRIMARY OUTCOMES:
Change in Social Support | intervals of 1, 2, 3, and 6 months post-baseline assessment
  Participants will complete the 5-item Social Support subscale of the Assessment of Recovery Capital (ARC) to assess social support. The difference between the post-baseline and baseline measures will be assessed.
Change in Financial Barriers to SUD Recovery | intervals of 1, 2, 3, and 6 months post-baseline assessment
  These barriers include lack of stable housing, transportation, and cost of recovery services. Participants will complete the Housing and Safety Subscale of the Assessment of Recovery Capital (ARC) to assess social support and housing stability. The difference between the post-baseline and baseline measures will be assessed.
Change in Situational Barriers to SUD Recovery | intervals of 1, 2, 3, and 6 months post-baseline assessment
  The barriers measured will be (1) long delays for treatment, (2) complexity of navigating the healthcare system, (3) lack of programs in one's community, (4)lack of professional help, (4) and not knowing where to go for help. The response options are binary (yes, they think this is a barrier to their recovery', or 'no, not a barrier to recovery'). Responses to these questions (0=no, 1=yes) will be summed to determine situational barriers. The difference between the post-baseline and baseline measures will be assessed.
Change in Inhibitory Control | baseline and 6 months post-baseline assessment
  Inhibitory control will be assessed behaviorally using a 150 - 200 trial computerized 'Stop Signal' Task, the most common measure of this construct. Stop Signal Reaction Time (SSRT) and Stop trial accuracy will be measured and compared across time points.
Change in Resting State EEG beta poewer | baseline and 6 months post-baseline assessment
  We will measure both absolute and relative powers for beta (14-25 Hz) bands using a 24-channel Soterix Medical EEG.
Change in Striatal Dopaminergic Functioning | baseline and 6 months post-baseline assessment
  Consistent with previous research, we will assess average spontaneous eyeblink rate, a well-validated indirect proxy for available levels of striatal tonic dopamine.
Change in Risk-Taking | baseline and 6 months post-baseline assessment
  Risk-taking will be measured using the 7-item Risk Propensity Scale (Meertens & Lion, 2008). Higher scores on this scale indicate greater risk-taking propensity.
Change in Emotion Regulation | baseline and 6 months post-baseline assessment
  The Emotion Regulation Questionnaire (ERQ-10) will be used to assess these emotion regulation strategies and skills.
Change in Goal-Related Activities | baseline and 6 months post-baseline assessment
  Participants will complete the 5-item Meaningful Activities from the Assessment of Recovery Capital questionnaire. The 5 items will be summed for a total score.

SECONDARY OUTCOMES:
Engagement in Recovery Services | intervals of 1, 2, 3, and 6 months post-baseline assessment
  Active involvement in recovery programs. This is a binary response question. Participants are asked "Are you actively involved in a recovery program right now?". Response options are 'yes' or 'no'. We will measure the change over time in engagement for each participant and compare the percentage of those in the intervention and control arm that are actively involved in recovery services at each time point.
Hospital Visit Frequency | six months pre- and post-baseline assessment
  number of readmissions and number of emergency department visits
Substance Use Severity | intervals of 1, 2, 3, and 6 months post-baseline assessment
  Frequency of substance use in past 30 days measured using the Addiction Severity Index (ASI-Lite).
Emotional Well-being | intervals of 1, 2, 3, and 6 months post-baseline assessment
  Participants will be asked to self-report two items about their emotion well-being on a scale of 0 (Not at all) to 9 (Severely). The questions are "In the past 30 days, how much have you been bothered by feeling sad, down, or uninterested in life?" and "In the past 30-days, have you felt anxious or nervous?".
Life Satisfaction | intervals of 1, 2, 3, and 6 months post-baseline assessment
  Participants will be asked to self-report their life satisfaction using a single item question on a scale of 1 (Very Satisfied) to 4 (Very Dissatisfied). Change across time on this scale will be measured.

CONTACTS AND LOCATIONS:
Locations (1):
- Greenville Memorial Hospital, Greenville, South Carolina, United States

REFERENCES:
- [Derived] Cupp JA, Byrne KA, Herbert K, Roth PJ. Acute Care Utilization After Recovery Coaching Linkage During Substance-Related Inpatient Admission: Results of Two Randomized Controlled Trials. J Gen Intern Med. 2022 Aug;37(11):2768-2776. doi: 10.1007/s11606-021-07360-w. Epub 2022 Mar 16. PMID 35296984